CLINICAL TRIAL: NCT01962519
Title: A Randomized Clinical Trial of Early Oral Feeding as a Component of Accelerated Recovery Protocol After Total Gastrectomy for Cancer
Brief Title: Early Oral Feeding After Total Gastrectomy for Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Marek Sierzega, Dr, Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: K/ZDS/002306; K/ZDS/002306 (Other: Jagiellonian University)
Record Dates: First submitted 2013-10-09; First posted 2013-10-14 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-10

CONDITIONS: Adenocarcinoma of the Stomach
Keywords: gastrectomy; gastric cancer; oral feeding; complications
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early oral feeding (Experimental): Early oral feeding starting with liquids on postoperative day (POD) 1, followed by a soft diet on POD 2, and solid foods on day 3
  Interventions: Dietary Supplement: Early oral feeding
- Delayed oral feeding (No Intervention): Delayed oral feeding starting with liquids on postoperative day (POD) 4, followed by a soft diet on POD 5, and solid foods on day 6

INTERVENTIONS:
Dietary Supplement: Early oral feeding — Oral fluids starting on POD 1, followed by a soft diet (thin purée six times a day) on day 2, and regular solid diet thereafter
  Arms: Early oral feeding

SUMMARY:
The aim of this study is to evaluate the possibility of shortening postoperative hospital stay after gastrectomy by early oral feeding as a component of an enhanced recovery protocol (ERAS).

ELIGIBILITY:
Inclusion Criteria:

* Total gastrectomy for cancer
* Age 18 - 80 years
* Informed consent

Exclusion Criteria:

* Numerous hepatic and peritoneal metastases
* Extended resections (pancreas, colon)
* Preoperative malnutrition requiring total parenteral nutrition
* Emergency surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative hospital stay | Participants will be followed for the duration of hospital stay, an expected average of 8 days
  Time between surgery and patient discharge

SECONDARY OUTCOMES:
Morbidity | Participants will be followed for the duration of hospital stay, an expected average of 8 days
  Any complication occurring during hospital stay

OTHER OUTCOMES:
Re-admissions | 30 days after discharge
  Hospital readmissions within 30 days after discharge
Effective oral feeding | Participants will be followed for the duration of hospital stay, an expected average of 8 days
  Time to reach oral feeding covering 75% of patient's requirements
Quality of life | Preoperatively, postoperative day 7, 14 days after discharge
  Quality of life measured by EORTC QLQ-C30 and EORTC QLQ - STO22
Laboratory parameters | Preoperatively, postoperative day 1 and 8
  Laboratory tests, including lymphocyte count, blood albumin, blood prealbumin

CONTACTS AND LOCATIONS:
Overall Officials: Jan Kulig, prof., Study Chair — First Department of Surgery, Jagiellonian University Medical College, Krakow, Poland
Locations (1):
- First Department of Surgery, Jagiellonian University Medical College, Krakow, Malopolska, Poland